CLINICAL TRIAL: NCT05381025
Title: The Effect of Oral Kavalactones on Sleep and Cortisol in a Cohort of Healthy Adult Males Preparing for Military Special Forces Training
Brief Title: Kavalactones on Sleep and Cortisol in Healthy Special Forces Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thorne HealthTech, Inc (Industry)
Collaborators: Performance First (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: THT002-PFKV01
Record Dates: First submitted 2022-05-09; First posted 2022-05-19 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Sleep
Keywords: Sleep; Kava; Piper methysticum; Stress; Cortisol; Special Operations

STUDY DESIGN:
Intervention Model Description: Participants will be divided into two arms which will cross-over during a washout period such that each participant will take the active and the placebo in one phase of the two-phase study.
Who Masked: Participant, Investigator
Masking Description: Participants will be aware of the contents of the active material but will not be informed as to whether they will begin or end the study with the active vs the placebo. Study Managers will also not be aware of what an individual participant is taking during the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active to Placebo (Cohort 1) (Experimental): Participants randomly allocated to Cohort 1 for Phase 1 will begin the study taking the active ingredient and will cross-over to taking placebo in Phase 2 of the study after a washout period.
  Interventions: Dietary Supplement: Kava (Piper methysticum) extract
- Placebo to Active (Cohort 2) (Experimental): Participants randomly allocated to Cohort 2 for Phase 1 will begin the study taking the placebo and will cross-over to taking the active ingredient in Phase 2 of the study after a washout period.
  Interventions: Dietary Supplement: Kava (Piper methysticum) extract

INTERVENTIONS:
Dietary Supplement: Kava (Piper methysticum) extract — Each dose (3 capsules) contains kavalactones (225 mg) and silicified microcrystalline cellulose.

SUMMARY:
This research study is being done to better understand the effects of kava supplementation on sleep quality and salivary cortisol in the context of the acute physical and psychological stress of military special forces preparation training. Kava is a botanical dietary supplement derived from the plant Piper methysticum. Cortisol is a hormone associated with stress.

DETAILED DESCRIPTION:
Acute physical and behavioral stress can interfere with sleep quality and cause cortisol to increase. This can have a negative impact on quality of life and the ability to perform optimally.

Kava, derived from the rootstumps of the Piper methysticum plant, has been utilized traditionally, socially, and for its calmative properties by the peoples of Oceania for millennia. Kava has been available as a dietary supplement for decades.

Participants in this placebo-controlled cross-over study will be enrolled concurrently with a special operations prep class during which they will be experiencing significant physical and mental stressors. Participants will be divided into two arms - one taking kava and the other taking placebo for the first two-week phase of the study. Following a washout and cross-over, participants will switch what they are taking for the second two-week phase.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Provides consent to participate in the study
* Understands and agrees to follow all study procedures and limitations

Exclusion Criteria:

* Female
* Use of kava within the past 8 weeks
* Use of over the counter or prescription sleep aids including dietary supplements within the past 8 weeks
* Use of acetaminophen that cannot be discontinued or replaced with an NSAID during the study
* Known liver disease or dysfunction
* Known kidney disease or dysfunction
* Any prior adverse reaction or known sensitivity or allergy to kava or related botanicals (peppers)
* Recent history of clinical depression or anxiety diagnosis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-10-09 (Actual)

PRIMARY OUTCOMES:
Change in Salivary Cortisol - Phase 1 | Day 1 and 15
  Diurnal salivary samples will be collected and tested for cortisol levels [ng/ml].
Change in Salivary Cortisol - Phase 2 | Day 1 and 15
  Diurnal salivary samples will be collected and tested for cortisol levels [ng/ml].
Change in Sleep Latency, Duration, and Quality - Phase 1 | Day 1, 8, and 15
  Data from the Restorative Sleep Questionnaire-Weekly (RSQ-W) [Total score 0-100; higher indicates better restorative sleep] plus other selected sleep questions will be combined to assess participant sleep during the study.
Change in Sleep Latency, Duration, and Quality - Phase 2 | Day 1, 8, and 15
  Data from the Restorative Sleep Questionnaire-Weekly (RSQ-W) [Total score 0-100; higher indicates better restorative sleep] plus other selected sleep questions will be combined to assess participant sleep during the study.

SECONDARY OUTCOMES:
Change in General Mood - Phase 1 | Day 1, 8, and 15
  Data from the Depression, Anxiety, and Stress Scale-21 (DASS-21) [Total score 0-63; higher is more distressed] will be used non-diagnostically to generate comparative scores which will be analyzed against the cortisol findings to assist in the interpretation of the kava-related outcomes.
Change in General Mood - Phase 2 | Day 1, 8, and 15
  Data from the Depression, Anxiety, and Stress Scale-21 (DASS-21) [Total score 0-63; higher is more distressed] will be used non-diagnostically to generate comparative scores which will be analyzed against the cortisol findings to assist in the interpretation of the kava-related outcomes.
Change in Motivation and Volition - Phase 1 | Day 1, 8, and 15
  Data from the Cravings for Rest and Volitional Energy Expenditure Scale (CRAVE) [Total score 0-50; higher is more motivated] will be used to assess participant motivation to perform in the context of the strenuous and demanding training schedule of this Prep Class.
Change in Motivation and Volition - Phase 2 | Day 1, 8, and 15
  Data from the Cravings for Rest and Volitional Energy Expenditure Scale (CRAVE) [Total score 0-50; higher is more motivated] will be used to assess participant motivation to perform in the context of the strenuous and demanding training schedule of this Prep Class.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Schmidt, PhD, MPhil, Principal Investigator — Advanced Pattern Analysis & Countermeasures Group
Locations (1):
- Performance First, Virginia Beach, Virginia, United States

IPD SHARING:
Plan to Share IPD: No